CLINICAL TRIAL: NCT05933668
Title: Phase I Clinical Study of YK0901 Injection for the Treatment of Advanced Solid Tumors With HLA-A * 11:01 Positive and KRAS G12V Mutation
Brief Title: Mutant KRAS G12V-specific TCR Transduced T Cell Therapy for Advanced Solid Tumor
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Yingkai Saiwei（Beijing）Biotechnology Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YK0901
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YK0901 cells (Experimental): Patients will undergo lymphocytapheresis, then treatment with TCR-T cells (at escalating doses) + IL-2.Accelerated titration and "3 + 3" dose escalation were used in this trial . Five dose levels were set up: the dose level was 1: 1× 108 ± 20%（8×107~1.2×108）; the dose level was 2: 1 × 109 （±20%：8×108~1.2×109）; the dose level was 3: 5 × 109 （±20%：4×109~6×109）; the dose level was 4: 2 × 1010 （±20%：1.6×1010~2.4×1010）; the dose level was 5: 5 × 1010 （±20%：4×1010~6×1010）.
  Interventions: Biological: YK0901 cells

INTERVENTIONS:
Biological: YK0901 cells — On day 0, the TCR-T cells will be administered one time. Drug: Fludarabine + Cyclophosphamide+Oxaliplatin Fludarabine: 25mg/m²/day×3days Cyclophosphamide: 300mg/m²/day×3 days Oxaliplatin：100mg×1day Drug: IL-2 After 18-24 hours of infusion of YK0901 cells, the patients will be given a small dose of IL-2 subcutaneously, 500,000 IU/time, twice a day (interval 10-12 hours), for 14 days.

SUMMARY:
This study is a single center, open, single arm, dose increasing early clinical study. The purpose of this study is to evaluate the safety and efficacy of YK0901 immunotherapy in the treatment of patients with advanced solid tumor whose tumor antigen KRAS G12V expression is positive (HLA-A * 11:01).

DETAILED DESCRIPTION:
KRAS mutations exist in various cancers, especially pancreatic, lung and colorectal cancer. G12V is one of the most common mutation types for KRAS. It's challenging to chemically acquire the targeted drug for this mutation. Recent studies reported that this mutation peptides can form a neoepitope for T cell recognition.Our study aims to evaluate the safety and tolerability of YK0901 TCR-T cell for KRAS G12V positive advanced solid tumors.In this trial, 11 subjects with KRAS G12V mutations and matching HLA-A*11:01 subtypes are recruited for autologous TCR-T therapy.Within 1-7days after pretreatment, subjects will receive a single TCR-T infusion with an infusion dose of about 1×108～5×1010.Once every 12 hours within 24 hours after TCR-T cell infusion, recombinant human interleukin-2 will be injected intravenously for 14 days .

ELIGIBILITY:
Inclusion Criteria:

1.Age ≥18 years and ≤75 years. 2.Failure on or intolerance to systemic therapy for unresectable advanced cancer.

3.Patients must have at least one measurable lesion defined by RECIST 1.1. 4.Genotype and tumor antigen screening must meet the following two criteria: 1) HLA-A * 11:01 positive; 2) KRAS G12V positive 5.ECOG score 0-1 and expected survival time ≥3 months 6.Patients must meet the following criteria at screening and before preconditioning (baseline). If any laboratory test result is abnormal referring to the following criteria, it is acceptable to test one more time within 1week. If the test result is still abnormal, the patient is screen failed:

1. Hematology (no intensive blood transfusion (≥2 times within 1week), platelet transfusion or cell growth factor (except for recombinant erythropoietin) performed within 7days before the test): neutrophils (NE) ≥1.5×109 per liter, lymphocytes (LY) ≥0.5×109per liter (except for before preconditioning), platelets (PLT) ≥75×109per liter and hemoglobin (Hb) ≥8.0 g/dL.
2. Blood chemistry: creatinine clearance ≥mL/min, alanine aminotransferase (ALT) ≤2.5×ULN, aspartate aminotransferase (AST) ≤2.5×ULN, total bilirubin (TB) ≤2×ULN, serum lipase and amylase <1.5 ULN, alkaline phosphatase (ALP) ≤2.5 ULN; for patients with bone or hepatic metastasis, AST, ALT and ALP <5ULN.
3. Prothrombin time ≤ULN+4 seconds. 7.Women of childbearing potential must have negative serum pregnancy test result at screening and before preconditioning and agree to use an effective and reliable contraceptive method for at least 1 year after the last study treatment. Te acceptable methods include bilateral tubal ligation/bilateral salpingectomy or bilateral tubal occlusion; any approved oral, injection or implantation of hormone; or barrier contraceptive method: condoms containing spermicidal foam/gel/film/paste /suppositories or occlusive cap (diaphragm or cervical/fornix cap).

8.Voluntarily willing to participate in the study and sign the written informed consent.

9.No systemic anti-tumor therapy received within 2 weeks prior to peripheral blood mononuclear cell (PBMC) collection.

10.Blood oxygen saturation (finger oxygen detection)≥ 95% in a calm and non oxygenated state.

Exclusion Criteria:

1. Pregnant or lactating women.
2. HIV, treponema pallidum or HCV serology is positive.
3. Patients with any uncontrolled active infection, including, but not limited to, active tuberculosis or HBV infection (HBsAg positive or HBV DNA positive).
4. Patients with AEs induced by previous treatment that have not recovered to Common Terminology Criteria for Adverse Events (CTCAE) ≤1, except for alopecia and other tolerable events judged by the investigator or permitted laboratory abnormalities according to the protocol.
5. Patient allergic or intolerant to preconditioning drugs, including, but not limited to, fudarabine and cyclophosphamide or oxaliplatin; allergic to the components of YK0901; penicillin allergy history confrmed by positive skin test; or any severe allergy history-for example, anaphylactic shock.
6. Patients who have a history of organ transplantation or are waiting for organ transplantation.
7. Patients who have undergone major surgery or severe trauma within 4weeks before apheresis .
8. Patients with other serious diseases that may restrict them from participating in this study, such as poorly controlled diabetes (glycosylated hemoglobin HbA1c >8% undertreatment), poorly controlled hypertension judged by the investigator (blood pressure >160mmHg/100mmHg), severe cardiac insufficiency (left ventricular ejection fraction <50%), myocardial infarction or unstable arrhythmia or unstable angina pectoris, pulmonary embolism, chronic obstructive pulmonary disease, interstitial lung disease or clinically significant lung function test abnormalities in the past 6months.
9. Before apheresis and preconditioning, patients who have the following conditions, including, but not limited to: new-onset arrhythmia that cannot be controlled by medications; hypotension that requires the use of vasopressors; or bacterial, fungal or viral infections that require intravenous antibiotic, antiviral or antifungal treatment, and the investigator judged that they are not suitable to continue the experiment. Patients who use antibiotics to prevent infection can continue the study upon the judgment of the investigator
10. Patients who are expected to continue using immunosuppressive therapy during the trial (excluding physiological replacement therapy with glucocorticoids, such as prednisone<10mg/d or equivalent doses)
11. Patients with central nervous metastases.
12. Patients who have participated in other intervention clinical trials within 2 weeks.
13. Patients with adverse drug addiction or a history of drug abuse.
14. Patient with other malignant tumors within the past 2 years or at the present, except for cervical cancer in situ and basal cell carcinoma of the skin.
15. Patients who are unable or unwilling to comply with the clinical protocol, by the investigator's judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 2 years
Treatment related AEs | 2 years

SECONDARY OUTCOMES:
Antitumor efficacy-Objective response rate (ORR) | 2 years
  The number of cases in which tumor size is reduced to PR or CR / the total number of evaluable cases (%).
Antitumor efficacy-Progression-free survival (PFS) | 2 years
  The period from the day when the subject receives the infusion of cells to the first recorded tumor progression (whether treated or not) or death of any cause, which occurs first.
Antitumor efficacy-Overall survival (OS) | 2 years
  The period from the first infusion to any cause of death
Antitumor efficacy-Duration of response (DOR) | 2 years
  The period from the first evaluation of CR or PR to the first evaluation of PD or death of any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Department of GI Oncology, Peking University Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No